CLINICAL TRIAL: NCT00556764
Title: Development of Cognitive Assessment Tools in Parkinson Disease
Acronym: ANAM
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Institute for Neurodegenerative Disorders (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency); University of Oklahoma (Other)
Responsible Party: Principal Investigator, Danna Jennings, MD, Principal Investigator, Institute for Neurodegenerative Disorders
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: ANAM-PD-02; #76,160 (Other: IND Number)
Record Dates: First submitted 2007-11-08; First posted 2007-11-12 (Estimated); Last update posted 2012-02-09 (Estimated); Status verified 2012-02

CONDITIONS: Parkinson Disease
Keywords: ANAM; Parkinson's
MeSH Terms: conditions — Parkinson Disease | interventions — Iodine-123; Functional Neuroimaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 2 cohorts (Experimental): In this observational study 2 cohorts will participate. Cohort 1 will include people with Parkinson disease and Cohort 2 will include healthy volunteers.
  A subset of twelve subjects (8 PD and 4 HC) will be enrolled in the [123I] IBVM and SPECT imaging portion of this study
  Interventions: Drug: [123I] IBVM and SPECT imaging; Drug: Subjects will undergo the 123-I IBVM imaging visit

INTERVENTIONS:
Drug: [123I] IBVM and SPECT imaging — Subjects will be injected with up to 4 mCi of 123-I IBVM followed by SPECT imaging.
  Other Names: FUNCTIONAL BRAIN IMAGING
Drug: Subjects will undergo the 123-I IBVM imaging visit — Subjects will be injected with a bolus of up to 4 mCi of 123-I IBVM followed by serial SPECT imaging.
  Other Names: FUNCTIONAL BRAIN IMAGING

SUMMARY:
The main objectives of this protocol are as follows:

1. To assess the sensitivity and specificity of ANAM-PD in detecting cognitive status in patients with Parkinson disease (PD) and healthy controls (HC).
2. To validate the specific individual domains of the ANAM-PD cognitive battery by comparisons to available standardized cognitive evaluation scales administered to the patients with Parkinson disease with and healthy control subjects.
3. To evaluate the reliability of the ANAM-PD battery of tests by comparing repeated administrations of the ANAM-PD battery on a sub-set of subjects with Parkinson disease and healthy controls.
4. To characterize cholinergic neurotransmission through imaging the vesicular acetylcholine transporter binding with 123Iodobenzovesamicol (IBVM) and SPECT in PD patients and healthy controls.

DETAILED DESCRIPTION:
General Design and Methods The overall goal of this proposal is to validate ANAM-PD as an assessment tool for cognitive status in PD. We propose a comprehensive strategy to evaluate the sensitivity and specificity of ANAM-PD in detecting cognitive changes in patients with a diagnosis of PD (n=50) and healthy controls (n=25). The specific testing domains of the ANAM-PD battery will be validated against standardized neuropsychological testing, described in detail below. The reliability of the ANAM-PD battery will be evaluated through a test-retest procedure in a subset of 50 subjects (25 PD and 25 HC). This strategy will enable us to evaluate the individual domains of the ANAM-PD computerized cognitive test and establish a battery as a standard test to efficiently measure cognitive changes in PD. We also propose to explore functional neuroimaging of the cholinergic system using [123I] IBVM and SPECT, a marker of vesicular acetylcholine transporter and a measure of the integrity of the cholinergic neuronal system. Identifying and validating ANAM-PD as an efficient tool for assessing cognitive changes in PD and exploring the cholinergic transporter system in PD through functional neuroimaging could predict sub-sets of PD patients 'at risk' for developing dementia and help elucidate the neurochemistry related to cognitive decline in PD

ELIGIBILITY:
Inclusion and Exclusion Criteria

PD subjects

Inclusion criteria:

* The participant is 30 years or older.
* Written informed consent is obtained.
* Participants have a clinical diagnosis of Parkinson's disease based on Brain Bank Criteria.
* Mini-mental status examination (MMSE) score ≥24 or significant cognitive dysfunction based clinical mental status exam.
* Geriatric Depression Scales (GDS) ≤ 10.
* For females, non-child bearing potential a negative urine or serum pregnancy test on day of 123-I IBVM injection.

Exclusion criteria:

* The subject has a clinically significant abnormal laboratory value and/or clinically significant unstable medical or psychiatric illness
* The subject has any disorder that may interfere with drug absorption distribution, metabolism, or excretion (including gastrointestinal surgery).
* Pregnancy

Healthy Control Subjects

Inclusion criteria:

* The participant is 50 years or older.
* Written informed consent is obtained.
* Negative history of neurological or psychiatric illness based on evaluation by a research physician.
* Mini-Mental Status Exam score ≥28.
* For females, non-child bearing potential a negative urine or serum pregnancy test on day of 123-I IBVM injection.

Exclusion criteria:

* The subject has a clinically significant abnormal laboratory value and/or clinically significant unstable medical or psychiatric illness.
* The subject has any disorder that may interfere with drug absorption distribution, metabolism, or excretion (including gastrointestinal surgery).
* The subject has received an investigational drug within 60 days before the screening visit.

Min Age: 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2007-07; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
The overall goal of this proposal is to validate ANAM-PD as an assessment tool for cognitive status in PD | 6 mos

CONTACTS AND LOCATIONS:
Overall Officials: Danna L Jennings, MD, Principal Investigator — Institute for Neurodegenerative Disorders
Locations (1):
- Institute for Neurodegenerative Disorders, New Haven, Connecticut, United States

REFERENCES:
- [Background] Kabat MH, Kane RL, Jefferson AL, DiPino RK. Construct validity of selected Automated Neuropsychological Assessment Metrics (ANAM) battery measures. Clin Neuropsychol. 2001 Dec;15(4):498-507. doi: 10.1076/clin.15.4.498.1882. PMID 11935451